CLINICAL TRIAL: NCT03381001
Title: Influence of Post-thaw Embryo Culture Interval Before Embryo Transfer on Assisted Reproduction Success Rates
Brief Title: Influence of Post-thaw Embryo Culture Interval on Assisted Reproduction Success Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Selmo Geber, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEC+1
Record Dates: First submitted 2017-12-11; First posted 2017-12-21 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Infertility
Keywords: cryopreservation; human embryos; vitrification; embryo culture; embryo transfer; pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Culture Techniques; Embryo Transfer

STUDY DESIGN:
Intervention Model Description: prospective, randomized, triple-blinded study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- embryo transfer after embryo thaw (Active Comparator): Embryos will be transferred at the same day of the thawing procedure
  Interventions: Procedure: embryo transfer with no culture
- embryo transfer after thaw and culture (Experimental): Embryos will be transferred one day after thawing procedure
  Interventions: Procedure: embryo transfer after thaw and culture

INTERVENTIONS:
Procedure: embryo transfer after thaw and culture — embryos will be kept in culture after thawing for one day before transfer for the uterus
  Arms: embryo transfer after thaw and culture
Procedure: embryo transfer with no culture — embryos will be transfer with no culture after thaw
  Arms: embryo transfer after embryo thaw

SUMMARY:
The transfer of frozen / thawed embryos has been routinely performed in the last 30 years as part of Assisted Reproduction treatment (ART). Currently, more than 50% of couples submitted to ART have surplus embryos eligible for freezing followed by transfer in subsequent cycles. Therefore the selection criteria for the thawed embryos to be transferred must be rigorous in order to maximize pregnancy and of live birth rates. Usually, the evaluation of the embryos before transfer can be performed based on blastomeres survival after a short culture period between thaw and embryos transfer, i.e., 2 to 5 hours, or based on embryo development over a prolonged period of culture (18h to 24h). Post-thaw embryo culture might have an impact on the recovery of mitosis and normal cellular functions. However, until now, there is no consensus in the literature on which post-thaw culture interval has a better impact on pregnancy and live birth rates. Also, blastocysts formation after freezing/thawing of embryos at cleavage stage may bring relevant information about post-thaw culture. Moreover, this strategy can be used as an alternative treatment. Therefore, the authors proposed this prospective randomized, triple-blind study to evaluate the impact of post-thaw embryo culture on the pregnancy and live birth rates.

ELIGIBILITY:
Inclusion Criteria:

* patients submitted to ART treatment due to infertility that had frozen embryos and need an embryo transfer after endometrial preparation and embryo thawing

Exclusion Criteria:

* patients that does not reach criteria for frozen embryo transfer (thin endometrium, bleeding, inappropriate use of hormones)
* difficult embryo transfer
* embryos that were frozen twice

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only women can have an embryo transfer
Enrollment: 268 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
pregnancy rates | 8 weeks
  percentage of patients that become pregnant after Frozen embryo transfer

SECONDARY OUTCOMES:
implantation rate | 6 weeks
  percentage of gestational sac according to the number of transferred embryos
embryo development | 24 hours
  percentage of embryos that develop after thawing and before transfer

CONTACTS AND LOCATIONS:
Overall Officials: selmo Geber, MD PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Hospital das Clinicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
we don't have permission to share participant data

REFERENCES:
- [Result] Roque M, Lattes K, Serra S, Sola I, Geber S, Carreras R, Checa MA. Fresh embryo transfer versus frozen embryo transfer in in vitro fertilization cycles: a systematic review and meta-analysis. Fertil Steril. 2013 Jan;99(1):156-162. doi: 10.1016/j.fertnstert.2012.09.003. Epub 2012 Oct 3. PMID 23040524
- [Result] Roque M, Valle M, Guimaraes F, Sampaio M, Geber S. Cost-Effectiveness of the Freeze-All Policy. JBRA Assist Reprod. 2015 Aug 1;19(3):125-30. doi: 10.5935/1518-0557.20150028. PMID 27203090
- [Result] Roque M, Valle M, Guimaraes F, Sampaio M, Geber S. Freeze-all policy: fresh vs. frozen-thawed embryo transfer. Fertil Steril. 2015 May;103(5):1190-3. doi: 10.1016/j.fertnstert.2015.01.045. Epub 2015 Mar 4. PMID 25747130
- [Result] Roque M, Valle M, Guimaraes F, Sampaio M, Geber S. Freeze-all cycle for all normal responders? J Assist Reprod Genet. 2017 Feb;34(2):179-185. doi: 10.1007/s10815-016-0834-x. Epub 2016 Nov 5. PMID 27817036
- [Result] Roque M, Valle M, Kostolias A, Sampaio M, Geber S. Freeze-all cycle in reproductive medicine: current perspectives. JBRA Assist Reprod. 2017 Feb 1;21(1):49-53. doi: 10.5935/1518-0557.20170012. PMID 28333033
- [Derived] Colodetti L, Pinho de Franca P, Sampaio M, Geber S. Do different culture intervals (2 x 24 hours) after thaw of cleavage stage embryos affect pregnancy rates? A randomized controlled trial. Cryobiology. 2020 Aug;95:80-83. doi: 10.1016/j.cryobiol.2020.06.002. Epub 2020 Jun 10. PMID 32533985